CLINICAL TRIAL: NCT04371510
Title: Blood Innate Biomarkers as Predictors of COVID-19 Disease Progression in Recently Infected Chronic Haemodialysis Patients
Brief Title: Blood Biomarkers as Predictors of COVID-19 Disease Progression in Recently Infected Chronic Haemodialysis Patients
Acronym: PredictCovid-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-PP-08
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 by SARS-CoV-2 Infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: PredictCOVID-D study. Covid-19 chronic haemodialysis patients with moderate symptoms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Covid-19 patients with moderate symptoms (Other): Whole blood, culture supernatant, serum
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — a blood sample is taken on Covid-19 chronic haemodialysis patients with moderate symptoms

SUMMARY:
SARS-CoV-2 induces over-production of inflammatory cytokines, and especially interleukin-6 (IL-6). The apparently strong association between blood levels of inflammaory cytokines and SARS-CoV-2 disease severity has led clinicians to evaluate the administration of steroids or anti-IL-6 antagonists in severely ill patients. As of this day, biomarkers capable of predicting clinical disease progression in Covid-19 patients with mild-to-moderate symptoms have not yet been formally identified. Identifying such markers and evaluating their predictive value may be exploited to guide patient care management, and as such forms the core objective of this proposal.

Because of strong inter-individual variations in the ability of innate immune cells to produce cytokines, the hypothesis the investigators formulate and intend to test is that innate IL-6 responsiveness varies between recently infected Covid-19 patients and could predict disease outcome.

To test this hypothesis, the investigators propose to follow recently infected chronic haemodialysis patients with moderate Covid-19 symptoms. These patients stand a higher risk to progress to severe disease. The investigators plan to collect a blood sample in these patients using a system whereby ex vivo cytokine production is initiated in the very same blood collection tube without prior separation and centrifugation, thus reducing labour and operator bias. After incubation with or without known innate immune stimuli, the cell-free phase from each collection-culture tube will be assayed for IL-6 content. Associations between IL-6 content and disease outcome (encephalopathy, transfer to acute care or death) will be determined in 115 Covid-19 chronic haemodialysis patients with moderate symptoms followed in 9 centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage chronic renal disease requiring haemodialysis support;
* SARS-CoV-2 positive (RT-PCR);
* COVID-19 symptoms at least once over a 8-day period preceding inclusion;
* Hospitalized or outpatients in one of the study centers: CHU de Nice, CHU de Strasbourg, Hôpital Necker (APHP), Hôpital Kremlin Bicêtre (APHP), Hôpital Pitié-Salpétriêre (APHP), Hospices Civils de Lyon, CHU de Saint-Etienne, CHU de Montpellier, Hôpital La Conception (APHM);
* Age > 18 years;
* Free and informed consent.

Exclusion Criteria:

* Age > 85 years ;
* Peritoneal dialysis;
* Onset of symptoms (fever and/or cough) for more than 8 days;
* Acute respiraytory distress despite oxygen therapy, 02 ≥ 4L/min, arterial pressure < 85/55 mmHg or hemodynamic instability at time of inclusion, encephalopathy with Glasgow coma scale < 14;
* Treatment with non-steroids anti-inflammatory agents within the laste 14 days preceding onset of symptoms;
* Active bacterial or fungal infection documented at inclusion;
* Pregnancy;
* Under guardianship or curatorship;
* Non-affiliated person with Social Security.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Predictive value of IL-6 contents of whole blood samples after ex vivo stimulation | 10 months
  Quantity of IL-6 in of whole blood samples after ex vivo co-stimulation with LPS and ATP in Covid-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: sicard antoine, ph, Principal Investigator — Néphrologie, CHU de Nice
Locations (1):
- CHU de nice, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided